CLINICAL TRIAL: NCT01606384
Title: A Double-blind, Placebo-controlled Study Evaluating the Pharmacodynamic Effects of Two Fixed Doses of SSR149415 (250 mg Bid and 100 mg Bid) on Hypothalamic-pituitary-adrenal Axis Function in Outpatients With Major Depressive Disorder
Brief Title: Evaluation of the Potential Effects of SSR149415 on the Hypothalamic-pituitary-adrenal Axis in Outpatients With Major Depressive Disorder
Acronym: NAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDY5467
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 1-(5-chloro-1-((2,4-dimethoxyphenyl)sulfonyl)-3-(2-methoxyphenyl)-2-oxo-2,3-dihydro-1H-indol-3-yl)-4-hydroxy-N,N-dimethyl-2-pyrrolidinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Twice daily
  Interventions: Drug: Placebo
- SSR149415 - 100mg (Experimental): Twice daily
  Interventions: Drug: VASOPRESSIN V1B RECEPTOR ANTAGONIST (SSR149415)
- SSR149415 - 250mg (Experimental): Twice daily
  Interventions: Drug: VASOPRESSIN V1B RECEPTOR ANTAGONIST (SSR149415)

INTERVENTIONS:
Drug: VASOPRESSIN V1B RECEPTOR ANTAGONIST (SSR149415) — Pharmaceutical form: Capsule Route of administration: oral
  Arms: SSR149415 - 100mg; SSR149415 - 250mg
Drug: Placebo — Pharmaceutical form: Capsule Route of administration: Oral
  Arms: Placebo

SUMMARY:
Primary Objective:

- To evaluate the effects of two fixed doses of SSR149415 (250 mg bid and 100 mg bid) on hypothalamic-pituitary-adrenal axis function in patients with major depressive disorder.

Secondary Objectives:

* To evaluate the tolerability and safety of SSR149415 in patients with major depressive disorder.
* To evaluate the efficacy of two fixed doses of SSR149415 compared to placebo in patients with major depressive disorder.
* To evaluate plasma concentrations of SSR149415.

DETAILED DESCRIPTION:
The study consisted of three segments (A, B and C). Segment A was a 1 to 4-week, drug-free, screening and baseline period. Segment B was a 4-week, double-blind period. After the last dose of double-blind study medication in Segment B, all patients had to enter Segment C, a 1-week drug-free, follow-up period.

The total study duration for one patient participating in all segments of the study was 6 weeks.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of major depressive disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition-Text Revision (DSM-IV-TR) and the Mini International Neuropsychiatric Interview (MINI) criteria.

Exclusion criteria:

* Outpatients unwilling to be hospitalized a total of 6 nights and 8 days.
* Total score of less than 21 (<21) on the 17-item Hamilton Depression Rating Scale (HAM-D) at Visit 1 (Day -7) or Visit 5 (Day -1).
* Patients whose current depressive episode is diagnosed with psychotic features, catatonic features, seasonal pattern or post-partum onset or is secondary to a general medical disorder.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months according to the MINI, except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Segment B: any antipsychotic within 3 months; fluoxetine within 1 month; any monoamine oxidase inhibitor (MAOI) within 2 weeks; any other antidepressant, anxiolytic, sedative-hypnotic, or mood-stabilizer (lithium, anticonvulsants) within 7 days except permitted concomitant medications
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Cortisol plasma concentration response to Corticotropin releasing factor (CRF) administration before and after 27 days of dosing | 4 weeks

SECONDARY OUTCOMES:
Adrenocorticotropic hormone (ACTH) plasma concentration response to CRF administration before and after 27 days of dosing | 4 weeks
Number of patients with adverse events | Up to 6 weeks
Changes in Hamilton Depression Rating Scale (HAM-D) depressed mood, factor and core items scores | Baseline, 4 weeks
Changes Clinical Global Impression (CGI) Severity and Improvement scores | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Griebel G, Beeske S, Stahl SM. The vasopressin V(1b) receptor antagonist SSR149415 in the treatment of major depressive and generalized anxiety disorders: results from 4 randomized, double-blind, placebo-controlled studies. J Clin Psychiatry. 2012 Nov;73(11):1403-11. doi: 10.4088/JCP.12m07804. Epub 2012 Oct 16. PMID 23146246